CLINICAL TRIAL: NCT02957812
Title: The Effects of 12-week Custom-made Orthotic Intervention on the Structure and Function of the Foot of Healthy Young Adults During Gait Termination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Katrina Protopapas, Principal Investigator, Wilfrid Laurier University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5114
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Flatfoot
Keywords: Gait; Balance Control; Orthotics
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orthotics (Experimental): Custom made orthotic provided for study
  Interventions: Device: Custom-made Foot Orthotics (CFO)
- Control (No Intervention): Wearing own footwear

INTERVENTIONS:
Device: Custom-made Foot Orthotics (CFO) — Provides longitudinal arch support
  Arms: Orthotics

SUMMARY:
The purpose of this study is to explore the long-term effects that orthotics imposes on the structure and function of the foot. The objectives of the study are to determine if the use of custom-made foot orthotics (CFO) cause: (a) changes to the structure of the plantar intrinsic muscles, (b) changes in the rate of muscle activity and timing in the plantar intrinsic muscles and (c) creates any changes in balance control during gait termination. The aim of the study is to enhance the appropriate dispensing of orthotics, and whether additional measures, such as rehabilitation exercises are necessary to increase their overall effectiveness in the clinical setting.

DETAILED DESCRIPTION:
Between 20-30 healthy young adults of both males and females will be recruited. A screening questionnaire will be administered to ensure that participants are appropriate for the study.

Once the participant has met the criteria of the study, the participants will be randomly allocated into one of two groups: (a) the control group or (b) the intervention group. Individuals that are selected to be in the intervention group, will be fitted with custom-made orthotics by an experienced pedorthist. The pedorthist will cast the foot posture using a foam impression to custom the design of the foot orthotic. The participant will have a week to acclimatize to the new environment, and if any discomfort arises the pedorthist will make any necessary corrections and the participant will have another week to acclimatize to the orthotic. The control group will not receive an intervention and ask to go about their daily life activities. All participants will undergo the same testing procedures at 6 and 12 weeks after baseline testing.

At baseline, 6 weeks and 12 weeks post-baseline, the researcher will take a diagnostic ultrasound image of the foot muscles prior to the gait trials. The researcher will also place 12 infrared markers and surface electrodes on the participant. All trials will be performed barefoot. The participants will then undergo a gait termination protocol. Participants will walk down an 8m walk-way with three force plates are embedded into the ground. Participants will be asked to walk to the end of the platform until instructed to stop. For 20% of the gait trials, the participants are walking forward until they hear an audio buzzer sound that will signal them to terminate their gait suddenly in the next two steps. All trials will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* a score of (+5) on the Foot Posture Index (FPI)
* navicular height < 3.6cm
* able to walk

Exclusion Criteria:

* have worn CFOs in the past year,
* current lower limb injury, leg or foot pain
* neurological or musculoskeletal disorders affecting the function of the foot
* previous history of lower limb surgery
* protein intake above the recommended daily allowance (RDA)
* medications that effect balance.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07-21 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Cross-sectional area (CSA) of intrinsic foot muscles | Baseline, 6 weeks, and 12 weeks post baseline
  the area of the cross section of a muscle perpendicular to its fibers
change in muscle activity and timing of Electromyography (EMG) | Baseline, 6 weeks, and 12 weeks
  muscle activity and muscle timing
change in Balance stability margin | Baseline, 6 weeks, and 12 weeks
  how close their body gets to perimeter of their base of support

SECONDARY OUTCOMES:
Range of motion (ROM) | Baseline and 12 weeks
  the degrees of motion that occurs at the joint
Stride Length | Baseline and 12 weeks
  the distance between heel strike of the same limb
Stride Width | Baseline and 12 weeks
  the lateral distance between midlines of each foot
Gait Velocity | Baseline and 12 weeks
  The rate of change in position with respect to time

CONTACTS AND LOCATIONS:
Locations (1):
- Biomechanics Lab, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided